CLINICAL TRIAL: NCT05796765
Title: A Phase 2B, Prospective, Double-Blind, Randomized Controlled Trial of the Micronized DHACM Injectable Product Compared to Saline Placebo Injection for the Treatment of Osteoarthritis of the Knee
Brief Title: Phase 2B Micronized DHACM vs. Saline in the Treatment of Knee Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued early by Sponsor
Sponsor: MiMedx Group, Inc. (Industry)
Collaborators: Rho, Inc. (Industry); United BioSource, LLC (Industry); NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIOA005
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. The injecting investigator(s) will not be blinded, but subjects and the evaluators performing safety and efficacy assessments will be blinded as to which treatment the subject received until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Micronized DHACM 40 mg (Experimental): Injection of 40 mg allogeneic micronized dehydrated human amnion chorion membrane (DHACM) suspended in 2.5 mL, 0.9% Sodium Chloride, USP
  Interventions: Biological: Micronized DHACM 40 mg
- Micronized DHACM 100 mg (Experimental): Injection of 100 mg allogeneic micronized dehydrated human amnion chorion membrane (DHACM) suspended in 2.5 mL, 0.9% Sodium Chloride, USP
  Interventions: Biological: Micronized DHACM 100 mg
- Saline (Placebo Comparator): Injection of 2.5 ml, 0.9% Sodium Chloride, USP
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Micronized DHACM 40 mg — Injection of 40 mg allogeneic micronized dehydrated human amnion chorion membrane (DHACM) suspended in 2.5 mL, 0.9% Sodium Chloride, USP
  Arms: Micronized DHACM 40 mg
Biological: Micronized DHACM 100 mg — Injection of 100 mg allogeneic micronized dehydrated human amnion chorion membrane (DHACM) suspended in 2.5 mL, 0.9% Sodium Chloride, USP
  Arms: Micronized DHACM 100 mg
Drug: Saline — Injection of 2.5 ml, 0.9% Sodium Chloride, USP
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the 40 mg and 100 mg doses of allogeneic micronized dehydrated human amnion/chorion membrane (micronized DHACM) injectable compared to 0.9% sodium chloride injection, placebo control for the treatment of knee osteoarthritis

DETAILED DESCRIPTION:
This is a phase 2B, prospective, double-blind, randomized controlled trial of the micronized DHACM injection as compared to saline placebo injection in the treatment of osteoarthritis of the knee. Approximately 30 experienced clinical centers in the United States and Denmark will participate in the study. Each subject will receive one injection and be evaluated for efficacy and safety during the 12-month observation period. Endpoints will be measured at 30 days, 60 days, 90 days, 120 days, 150 days, 180 days, 270 days and 365 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age ≥ 21 and ≤ 80 years.
2. Subject has a diagnosis of primary OA of the target knee (as per American College of Rheumatology clinical and radiological criteria) with OA symptoms (as reported by the subject) that have been present for at least 6 months prior to Screening.
3. Subject has Grade 2 or 3 OA of the target knee on the Kellgren Lawrence (KL) grading scale as evaluated by central reading of screening X-ray.
4. Subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study.
5. Subject must have a WOMAC pain score ≥ 4 and ≤ 9 out of 10 in target knee, at screening and baseline.
6. Subject must have tried and failed to adequately respond to 2 knee OA standard of care (SOC) therapies, including at least one pharmacological treatment, for a minimum of 3 months. SOC for knee OA include non-pharmacological (exercise, weight loss, knee braces, cane) and pharmacological treatments (topical nonsteroidal anti-inflammatory drugs [NSAIDs], oral NSAIDs, and intra-articular corticosteroids).
7. Subject must be willing to discontinue all current pain medications (including but not limited to oral, topical, intra-articular) during the duration of the study except for acetaminophen (paracetamol) which will be allowed as rescue, except as noted in inclusion criterion 10 below. Limited use of NSAIDS will be permitted at the discretion of the investigator for post injection pain only.
8. Subject must have a WOMAC pain subscale score in contralateral knee less than 4 out of 10, at screening and baseline visits.
9. Subject who is identified as having taking analgesics at their initial screening visit 1a must be willing to abstain from analgesics for a washout period of 5 half-lives of the analgesic plus 48 hours and return for screening visit 1b where WOMAC pain can be collected analgesic-free.
10. Subject must be willing to abstain from use of rescue medication (acetaminophen/paracetamol) for at least 72 hours prior to all study visits subsequent to screening.
11. For male subjects:

    1. Subject must agree to use highly effective contraception throughout the study.
    2. Subject must agree not to donate sperm during the study.
12. For female subjects:

    1. Subject is surgically sterile; or
    2. Has been amenorrheic for at least 1 year and is over the age of 55 years; or
    3. Has a negative urine pregnancy test and agrees to use acceptable contraceptive measures (e.g. hormonal contraceptives, barriers with spermicide, intrauterine device or vasectomized partner) from the time of informed consent through the end of the study; and
    4. Must commit to the use of highly effective form of birth control from the time of informed consent through the end of the study.
13. Subject must have vital signs within the following ranges at the screening visit and at the baseline visit before investigational product administration:

    1. Systolic blood pressure ≤140 and ≥90 mmHg,
    2. Diastolic blood pressure ≤90 and ≥60 mmHg,
    3. Heart rate <100 and >60 bpm,
    4. Temperature: normal,
    5. Respiratory rate <20 and >12 /min.

Exclusion Criteria:

1. Subject has Grade 1 or 4 OA of the target knee on the Kellgren Lawrence (KL) grading scale as evaluated by central reading of screening X-ray.
2. Subject has a BMI greater than 40 kg/m^2.
3. Subject has a clinical effusion (3+) of the target knee according to the Stroke Test grading system.
4. Subject has symptoms of locking, intermittent block to range of motion, or loose body sensation that could indicate meniscal displacement or an intra-articular loose body.
5. Subject has any active infection of the target knee, and/or any active systemic or local infection.
6. Subject has a history of allergy or sensitivity to any of the investigational product components, including aminoglycoside antibiotics.
7. Symptomatic pain in either or both hips that exceeds that of the target knee, as determined by investigator assessment.
8. Significant radicular back pain, as determined by investigator assessment.
9. Subject has rheumatoid arthritis, psoriatic arthritis, or has been diagnosed with any other disorder that is the primary source of their knee pain, including but not limited to: osteonecrosis, radiculopathy, bursitis, tendinitis, tumor, cancer.
10. Subject has documented history of gout or pseudogout.
11. Subject has fibromyalgia or any other chronic pain disorder.
12. Subject has an autoimmune disease or a known history of having acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV).
13. Subject has received any of the following to the target knee:

    1. Intra-articular hyaluronic acid (HA) injection within 24 weeks prior to screening;
    2. Intra-articular short-acting corticosteroid such as triamcinolone within 12 weeks prior; if long-acting (Zilretta) within 5 months prior to screening;
    3. Platelet rich plasma (PRP) injection within 6 months prior to screening;
    4. Is planning to receive physical therapy during the study;
    5. Has had or is planning to have major surgery or arthroscopy in the target knee within 52 weeks of treatment;
    6. History of a total knee arthroplasty.
14. Subject has a history of total knee arthroplasty in the contralateral knee within the last 12 months.
15. Subject has received any prior treatment with tissue engineered or amniotic products, including any MIMEDX product.
16. Subject has used an investigational drug, device, or biologic within 12 weeks or 5 half-lives of the investigational product prior to screening.
17. Subject has been exposed to investigational use of nerve growth factor (NGF) antagonists.
18. Subject uses any opioids to control their pain.
19. Subject is taking a drug with known or suspected immunosuppressive effects.
20. Subject with a history of systemic corticosteroid use within three months of screening and subjects who are likely to need systemic steroids during the study (e.g., poorly controlled asthma, severe COPD).
21. Subject is breast feeding.
22. Subject has had prior radiation therapy to the target or contralateral knee.
23. Subject is currently taking anticoagulant therapy (excluding Plavix or similar or low dose aspirin).
24. Subject has a known or suspected history of alcohol, narcotic or other drug abuse or substance dependence within the past 12 months, prior to screening.
25. Subject has any significant medical or psychiatric condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation.
26. Subject has any of the following uncontrolled co-morbid conditions: cirrhosis, Child Class B or C liver disease, or other clinically significant indicators of liver disease, such as portal hypertension; eGFR <60 mL/min/1.73 m^2 by the CKD-Epi formula; hemoglobin A1c >8.0 mmol/mol; hemoglobin <11.0 g/dL; coagulopathy; systolic blood pressure (BP) >140 or <90 mmHg, diastolic BP >90 or <60 mmHg, or heart rate (HR) ≥100 or ≤60 bpm.
27. Subject has a history of malignancy of any organ system (localized squamous or basal cell carcinoma of the skin are not exclusionary unless localized at the injection site), treated or untreated within 2 years of screening.
28. Subject has a worker's compensation or disability claim related to their knee osteoarthritis.
29. Subject requires more than intermittent use of a rollator, walker, cane, or other assistive devices.
30. Subject currently using marijuana in any form, including but not limited to topical or oral methods of use.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC pain subscale score between baseline and Day 180 | 180 days
  Efficacy Endpoint
Change in WOMAC function subscale score between baseline and Day 180 | 180 days
  Efficacy Endpoint
Proportions of subjects who report treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | 365 days
  Safety Endpoint

SECONDARY OUTCOMES:
Proportion of subjects who report greater than the minimal clinically important difference (MCID) improvement in WOMAC pain and function compared to baseline at Day 90 or Day 180 | 90 Days, 180 Days
  Secondary Efficacy Endpoint
Change in SF-36 physical component score (PCS), mental component score (MCS), and domain scores between baseline and Day 90 or Day 180 | 90 Days, 180 Days
  Secondary Efficacy Endpoint
Change in patient's global assessment (PtGA) of the target joint between baseline and Day 90 or Day 180 | 90 Days, 180 Days
  Secondary Efficacy Endpoint
Proportion of subjects who report greater than the minimal clinically important difference (MCID) improvement in patient's global assessment (PtGA) compared to baseline at Day 90 or Day 180 | 90 Days, 180 Days
  Secondary Efficacy Endpoint
Number of OMERACT-OARSI "Strict Responders" at Day 90 or Day 180 | 90 Days, 180 Days
  Secondary Efficacy Endpoint

OTHER OUTCOMES:
Proportion of subjects taking acetaminophen/paracetamol or any other non-study pain medication | 365 Days
  Exploratory Endpoint
Average amount (milligrams) of rescue medication used between Day 8 and Day 180 and between Day 180 and Day 365 | 180 Days, 365 Days
  Exploratory Endpoint
Time to initiation of use of acetaminophen/paracetamol or any other non-study pain medication, excluding the first 7 days following injection | 365 Days
  Exploratory Endpoint
Change in WOMAC pain subscale scores between baseline and additional time points | 30 Days, 60 Days, 90 Days, 120 Days, 150 Days, 270 Days, 365 Days
  Exploratory Endpoint
Change in WOMAC function subscale scores between baseline and additional time points | 30 Days, 60 Days, 90 Days, 120 Days, 150 Days, 270 Days, 365 Days
  Exploratory Endpoint

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Horizon Clinical Research, La Mesa, California
  - AppleMed Research Group, LLC, Miami, Florida
  - Health and Life Research Institute, LLC, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Premier Medical Associates, The Villages, Florida
  - Elite Clinical Trials, LLLP, Blackfoot, Idaho
  - Healthcare Research Network, Hazelwood, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - University Orthopedics Center - Altoona, Altoona, Pennsylvania
  - University Orthopedics Center - State College, State College, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - ClinRX Research Joseph, Inc., Carrollton, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah

IPD SHARING:
Plan to Share IPD: No